CLINICAL TRIAL: NCT03280303
Title: POLARIS: PALBOCICLIB IN HORMONE RECEPTOR POSITIVE ADVANCED BREAST CANCER: A PROSPECTIVE MULTICENTER NON-INTERVENTIONAL STUDY
Brief Title: Palbociclib in Real World Practice
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481082; POLARIS (Other: Alias Study Number)
Record Dates: First submitted 2017-09-01; First posted 2017-09-12 (Actual); Results first posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-05

CONDITIONS: Advanced Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- non-interventional study: This prospective, observational study will be conducted according to each site's routine clinical practice.
  Interventions: Other: non-interventional

INTERVENTIONS:
Other: non-interventional

SUMMARY:
This Non-Interventional Study will describe and analyze the clinical use of palbociclib in routine clinical practice in the treatment of advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥18 years or older.
2. Diagnosis of adenocarcinoma of the breast with evidence of metastatic disease or advanced disease not amenable to treatment with curative intent.
3. Documented HR+ (ER+ and/or PR+) tumor based on local standards.
4. Documented HER2- tumor based on local standards.
5. Physician has determined that treatment with palbociclib is indicated.
6. Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study.
7. Patients who in the opinion of the investigator are willing and able to comply with regular clinic visits as per standard of care practice at the site.

Exclusion Criteria:

1. Patients with a life expectancy of less than 3 months at the time of ABC diagnosis, per the investigator's judgment.
2. Patients participating in any interventional clinical trial that includes investigational or marketed products at the time of enrollment. (Patients participating in other investigator initiated research or NIS can be included as long as their standard of care is not altered by the study).
3. Patients on active treatment for malignancies other than ABC at the time of enrollment.
4. Patients who are unable to understand the nature of the study and are unwilling to sign an informed consent.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HR+/HER2- ABC patients whose treatment decision with palbociclib has been made by their treating physician and who meet the eligibility criteria will be invited to participate in the study.
Sampling Method: Probability Sample
Enrollment: 1285 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (292):
- United States (288):
  - Alabama Oncology, Alabaster, Alabama
  - Alabama Oncology, Bessemer, Alabama
  - Alabama Oncology, Birmingham, Alabama
  - Grandview Cancer Center, Alabama Oncology, Birmingham, Alabama
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Central Arkansas Radiation Therapy Institute, Little Rock, Arkansas
  - Central Arkansas Radiation Therapy Institute, Stuttgart, Arkansas
  - Sutter Auburn, Auburn, California
  - AIS Cancer Center at Adventist Health Bakersfield, Bakersfield, California
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Providence Health and Services Southern California, Burbank, California
  - Enloe Regional Cancer Center, Chico, California
  - John Muir Clinical Research Center, Concord, California
  - John Muir Medical Center, Concord Campus, Concord, California
  - Mount Diablo Solano Oncology Group, Concord, California
  - Global Cancer Research Institute, Inc., Gilroy, California
  - Breastlink Medical Group, Inc., Laguna Hills, California
  - Breastlink Medical Group, Inc., Newport Beach, California
  - Breastlink Medical Group, Inc., Orange, California
  - St. Jude Hospital Yorba Linda DBA St. Joseph Heritage Healthcare, Petaluma, California
  - Diablo Valley Oncology Hematology Medical Group, Pleasant Hill, California
  - Epic Care, Pleasant Hill, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Institute for Medical Research, Sacramento, California
  - Salinas Valley Medical Clinic Cancer Care, Salinas, California
  - Salinas Valley Memorial Healthcare System, Salinas, California
  - Santa Clara Valley Medical Center, San Jose, California
  - Cancer Research Collaboration/Breastlink Medical Group, Inc., Santa Ana, California
  - Ridley Tree Cancer Center, Santa Barbara, California
  - SANSUM Clinic, Santa Barbara, California
  - St. Jude Hospital Yorba Linda DBA St. Joseph Heritage Healthcare, Santa Rosa, California
  - Sansum Clinic, Solvang, California
  - St. Helena Hospital, St. Helena, California
  - St. Joseph's Medical Center, Stockton, California
  - Stockton Hematology Oncology Medical Group, Stockton, California
  - Cancer Treatment Center of Vacaville, Vacaville, California
  - Solano Hematology Oncology, Vallejo, California
  - Contra Costa Oncology, Walnut Creek, California
  - John Muir Medical Center, Walnut Creek Camous, Walnut Creek, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Boulder, Colorado
  - Rocky Mountain Cancer Centers, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Colorado West Healthcare System, dba Community Hospital, Grand Junction, Colorado
  - Colorado West Healthcare System, dba Grand Valley Oncology, Grand Junction, Colorado
  - Rocky Mountain Cancer Centers, Lakewood, Colorado
  - Rocky Mountain Cancer Centers, Littleton, Colorado
  - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers, Longmont, Colorado
  - Rocky Mountain Cancer Centers, Parker, Colorado
  - Rocky Mountain Cancer Centers, Pueblo, Colorado
  - Rocky Mountain Cancer Centers, Thornton, Colorado
  - Western Connecticut Health Network, Danbury, Connecticut
  - Western Connecticut Health Network, New Milford, Connecticut
  - Western Connecticut Health Network, Norwalk, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Cancer Research Institute, Boca Raton, Florida
  - Boca Raton Regional Hospital/Lynn Cancer Institute, Boca Raton, Florida
  - Cancer Specialists of North Florida, Fleming Island, Florida
  - Southeast Florida Hematology-Oncology Group, PA, Fort Lauderdale, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - University of Florida Health, Jacksonville, Florida
  - Cancer Specialists LLC, Jacksonville, Florida
  - Watson Clinic, Lakeland, Florida
  - Baptist Health Medical Group Oncology, LLC, Miami, Florida
  - Baptist Health Miami Cancer Institute, Miami, Florida
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - Cancer Specialists of North Florida - St. Vincent's Clay, Middleburg, Florida
  - Millennium Oncology Research Clinic/Hematology and Oncology Private Practice, Pembroke, Florida
  - Baptist Health Miami Cancer Institute, Plantation, Florida
  - Florida Cancer Research Institute, Plantation, Florida
  - Cancer Specialists of North Florida, Saint Augustine, Florida
  - Baptist Health Urgent Care Sawgrass, Sunrise, Florida
  - Northwest Georgia Oncology Centers, PC, Austell, Georgia
  - Northwest Georgia Oncology Centers, PC, Carrollton, Georgia
  - Northwest Georgia Oncology Centers, PC, Cartersville, Georgia
  - Northwest Georgia Oncology Centers, PC, Douglasville, Georgia
  - Gwinnett Hospital System, Inc. The Center for Cancer Care, Duluth, Georgia
  - Gwinnett Hospital System, Inc., Duluth, Georgia
  - Gwinnett Hospital System Inc., Lawrenceville, Georgia
  - Gwinnett Hospital System, Inc. The Center for Cancer Care, Lawrenceville, Georgia
  - Northwest Georgia Oncology Centers, PC, Marietta, Georgia
  - Northwest Georgia Oncology Centers, PC, Roswell, Georgia
  - Candler Medical Oncology Practice (CMOP)/Summit Cancer Care, Savannah, Georgia
  - Summit Cancer Care Research, Savannah, Georgia
  - Candler Medical Oncology Practice (CMOP), Savannah, Georgia
  - Gwinnett Hospital System, Inc. The Center for Cancer Care, Snellville, Georgia
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Presence St. Mary's Cancer Center, Bourbonnais, Illinois
  - Presence Saint Joseph Hospital, Chicago, Illinois
  - North Shore Oncology Hematology Associates, Crystal Lake, Illinois
  - North Shore Oncology-Hematology Associates, Crystal Lake, Illinois
  - Presence Infusion Care - Evanston, Evanston, Illinois
  - Joliet Oncology-Hematology Associates, LTD, Joliet, Illinois
  - Advocate Condell Medical Center, Libertyville, Illinois
  - North Shore Oncology-Hematology Associates, Libertyville, Illinois
  - Joliet Oncology-Hematology Associates, LTD, Morris, Illinois
  - Joliet Oncology-Hematology Associates, LTD, New Lenox, Illinois
  - Mid Illinois Hematology And Oncology Associates, Limited, Normal, Illinois
  - Quincy Medical Group, Quincy, Illinois
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - Presence Infusion Care - Skokie, Skokie, Illinois
  - Oncology Hematology Associates of Southwest Indiana, Newburgh, Indiana
  - McFarland Clinic, P.C., Ames, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Stormont Vail Regional Health Center, Topeka, Kansas
  - Stormont Vail Cotton O'Neill Cancer Center, Topeka, Kansas
  - University of Kansas Cancer Center, Westwood, Kansas
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Louisiana Hematology Oncology Associates, Baton Rouge, Louisiana
  - Our Lady of the Lake Regional Medical Center, Oncology 6, Baton Rouge, Louisiana
  - Pontchartrain Cancer Center, Covington, Louisiana
  - Pontchartrain Cancer Center, Hammond, Louisiana
  - Cancer Center at West Jefferson Medical Center, New Orleans Physician Services, Inc., Marrero, Louisiana
  - Crescent City Research Consortium, LLC, Marrero, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - Touro Infirmary, New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Maryland Oncology and Hematology, PA, Bethesda, Maryland
  - The Office of Frederick P. Smith, MD, Chevy Chase, Maryland
  - Maryland Oncology Hematology, P.A., Clinton, Maryland
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Maryland Oncology Hematology, P.A., Frederick, Maryland
  - Antietam Oncology and Hematology Group, PC, Haggerstown, Maryland
  - Maryland Oncology Hematology, P.A., Rockville, Maryland
  - Maryland Oncology Hematology, P.A., Silver Spring, Maryland
  - University of Maryland St. Joseph Medical Center, Towson, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - New England Hematology Oncology/Massachusetts General Cancer Center at Newton Wellesley Hospital, Newton, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Great Lakes Cancer Management, Grosse Pointe Woods, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Great Lakes Cancer Management, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology Hematology, PA, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fairview Southdale Medical Oncology Clinic, Edina, Minnesota
  - University of Minnesota Health Maple Grove Clinics, Maple Grove, Minnesota
  - Minnesota Oncology Hematology, PA, Minneapolis, Minnesota
  - Metro-Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Health Partners Institute, Saint Louis Park, Minnesota
  - Park Nicollet Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Minnesota Oncology Hematology, PA, Saint Paul, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA, Woodbury, Minnesota
  - North Mississippi Medical Center, Inc., Hematology and Oncology Research, Tupelo, Mississippi
  - Mercy Clinic St. Louis Cancer and Breast Institute, Ballwin, Missouri
  - St. Louis Cancer Care, LLP, Bridgeton, Missouri
  - St. Louis Cancer Care, LLP, Chesterfield, Missouri
  - Boone Hospital Center, Columbia, Missouri
  - Missouri Cancer Associates, Columbia, Missouri
  - St. Luke's Cancer Institute - East, Kansas City, Missouri
  - St. Luke's Cancer Institute, Kansas City, Missouri
  - St. Luke's Cancer Institute - Liberty, Liberty, Missouri
  - University of Kansas Cancer Center, North Kansas City, Missouri
  - Heartland Regional Medical Center/dba Cancer Care St. Joseph Mosaic Life Care, Saint Joseph, Missouri
  - Mercy Clinic St. Louis Cancer and Breast Institute, St Louis, Missouri
  - SSM Health St. Louis University Hospital, St Louis, Missouri
  - St. Louis University Cancer Center, St Louis, Missouri
  - St. Louis Cancer Care, LLP, St Louis, Missouri
  - Mercy Hospital St. Louis, St Louis, Missouri
  - Mercy Research - Mercy Heart Hospital St. Louis, St Louis, Missouri
  - Nebraska Hematology/Oncology, PC, Lincoln, Nebraska
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Hackensack University Medical Center, John Theurer Cancer Center, Hackensack, New Jersey
  - The Valley Hospital, Paramus, New Jersey
  - St. Luke's University Heatlh Network - Warren Hospital, Phillipsburg, New Jersey
  - CareMount Medical, Brewster, New York
  - New York Cancer and Blood Specialists, East Setauket, New York
  - CareMount Medical, Mount Kisco, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - New York Cancer and Blood Specialists, Patchogue, New York
  - New York Cancer and Blood Specialists, Port Jefferson Station, New York
  - New York Cancer and Blood Specialists, Riverhead, New York
  - New York Cancer and Blood Specialists, Smithtown, New York
  - White Plains Hospital, White Plains, New York
  - Asheville Hematology and Oncology, Asheville, North Carolina
  - Johnston Health Services Corporation - Clayton, Clayton, North Carolina
  - Haywood Infusion Center, Clyde, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - East Carolina University Brody School of Medicine, Greenville, North Carolina
  - DLP Maria Parham Medical Center, Henderson, North Carolina
  - Advent Health - Hendersonville, Hendersonville, North Carolina
  - University of North Carolina Regional Physicians Hematology Oncology, High Point, North Carolina
  - Novant Health Oncology Specialists, Kernersville, North Carolina
  - Duke Cancer Network, Laurinburg, North Carolina
  - Southeastern Regional Medical Center, Lumberton, North Carolina
  - Novant Health Oncology Specialists, Mount Airy, North Carolina
  - Novant Health Oncology Specialists, North Wilkesboro, North Carolina
  - Johnston Health Services Corporation - Smithfield, Smithfield, North Carolina
  - Novant Health Oncology Specialists, Statesville, North Carolina
  - Novant Health Oncology Specialists, Thomasville, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Hematology Oncology Associates, Inc., Canton, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Mid Ohio Oncology/Hematology, Inc. dba The Mark H. Zangmeister Center, Columbus, Ohio
  - Tri-County Hematology and Oncology Associates, Inc., Dover, Ohio
  - Tri-County Hematology and Oncology Associates, Inc., Massillon, Ohio
  - Mercy Health Perrysburg Cancer Center, Perrysburg, Ohio
  - Mercy Health St. Vincent Medical Center, Toledo, Ohio
  - Mercy Health Cancer Center, Toledo, Ohio
  - Mercy Health Youngstown dba St Joseph Warren Hospital, Warren, Ohio
  - Mercy Health Youngstown dba St. Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Northwest Cancer Specialists, PC, Portland, Oregon
  - Willamette Valley Cancer Institute and Research Center, Springfield, Oregon
  - St. Luke's University Health Network - Sacred Heart Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital - Allentown Campus, Allentown, Pennsylvania
  - St. Luke's Hematology Oncology Specialists, Bethlehem, Pennsylvania
  - St. Luke's University Heatlh Network, Bethlehem, Pennsylvania
  - St. Luke's University Heatlh Network, Easton, Pennsylvania
  - Pinnacle Health Cancer Center, Harrisburg, Pennsylvania
  - Pinnacle Health Cancer Institute, Harrisburg, Pennsylvania
  - Lancaster Cancer Center, Lancaster, Pennsylvania
  - Ortenzio Cancer Center at Pinnacle Health, Mechanicsburg, Pennsylvania
  - Charleston Cancer Center, Charleston, South Carolina
  - Greenville Health System, Easley, South Carolina
  - Tidelands Waccamaw Oncology/Georgrtown Hospital System, Georgetown, South Carolina
  - Greenville Health System, Greenville, South Carolina
  - Greenville Health System, Greer, South Carolina
  - Carolina Blood and Cancer Care Associates, PA, Lancaster, South Carolina
  - Tidelands Waccamaw Oncology/Georgrtown Hospital System, Murrells Inlet, South Carolina
  - Tidelands Waccamaw Oncology/Georgrtown Hospital System, Myrtle Beach, South Carolina
  - Carolina Blood and Cancer Care Associates, PA, Rock Hill, South Carolina
  - Greenville Health System, Seneca, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Greenville Health System, Spartanburg, South Carolina
  - M. Francisco Gonzalez, MD, PA, Sumter, South Carolina
  - Wellmont Bristol Regional Medical Center, Bristol, Tennessee
  - Wellmont Medical Associates Oncology and Hematology, Bristol, Tennessee
  - University of Tennessee/Erlanger Oncology and Hematology, Chattanooga, Tennessee
  - Wellmont Medical Associates Oncology and Hematology, Johnson City, Tennessee
  - Wellmont Cancer Institute, Kingsport, Tennessee
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Texas Oncology -Allen, Allen, Texas
  - Texas Oncology, Dallas, Texas
  - Texas Oncology-Denton South, Denton, Texas
  - Texas Oncology-El Paso Cancer Treatment Center, El Paso, Texas
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - Texas Oncology, Fort Worth, Texas
  - Texas Oncology - Southwest Fort Worth, Fort Worth, Texas
  - Texas Oncology, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University Medical Center Health System, Southwest Cancer Center, Lubbock, Texas
  - Texas Oncology, McAllen, Texas
  - Texas Oncology - McKinney, McKinney, Texas
  - Texas Oncology, Mesquite, Texas
  - Texas Oncology-Paris, Paris, Texas
  - Texas Oncology, Plano, Texas
  - Texas Oncology-San Antonio Downtown, San Antonio, Texas
  - Texas Oncology, San Antonio, Texas
  - Texas Oncology-San Antonio Stone Oak, San Antonio, Texas
  - Texas Oncology, Tyler, Texas
  - Virginia Cancer Specialists, Arlington, Virginia
  - Wellmont Medical Associates Oncology and Hematology, Bristol, Virginia
  - Cancer Specialists of Tidewater/Riverside Cancer Infusion Center, Chesapeake, Virginia
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Augusta Health Cancer Center, Fishersville, Virginia
  - Virginia Cancer Specialists, Gainesville, Virginia
  - Peninsula Cancer Institute/Riverside Cancer Infusion Center, Gloucester, Virginia
  - Virginia Cancer Specialists, Leesburg, Virginia
  - Bon Secours Memorial Regional Medical Center, Inc., Mechanicsville, Virginia
  - Bon Secours Richmond Community Hospital dba Oncology Associates at Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Cancer Institute @ St. Francis Medical Center, Midlothian, Virginia
  - Bon Secours Richmond Community Hospital dba Oncology Associates at St. Francis Medical Center, Midlothian, Virginia
  - Bon Secours St. Francis Medical Center, Inc., Midlothian, Virginia
  - Riverside Shore Cancer Center, Nassawadox, Virginia
  - Peninsula Cancer Institute/Riverside Cancer Infusion Center, Newport News, Virginia
  - Southwest Virginia Regional Cancer Center, Norton, Virginia
  - Delta Hematology/Oncology Associates, Portsmouth, Virginia
  - Bon Secours Richmond Community Hospital dba Oncologists Associates at St. Mary's Hospital, Richmond, Virginia
  - Bon Secours St. Mary's Hospital, Inc., Richmond, Virginia
  - Cancer Specialists of Tidewater/Riverside Cancer Infusion Center, Suffolk, Virginia
  - Cancer Specialists of Tidewater/Riverside Cancer Infusion Center, Virginia Beach, Virginia
  - Peninsula Cancer Institute/Riverside Cancer Infusion Center, Williamsburg, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Northwest Cancer Specialists, PC, Vancouver, Washington
  - West Virginia University Medicine - United Hospital Center, Bridgeport, West Virginia
  - Huntington Internal Medicine Group, Huntington, West Virginia
  - St. Mary's Medical Center, Huntington, West Virginia
  - West Virginia University, Mary Babb Randolph Cancer Center, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
- Canada (4):
  - Burnaby Hospital Cancer Centre, Burnaby, British Columbia
  - Trillium Health Partners, Mississauga, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Integrated University Center for Health and Social Services (CIUSSS) of Saguenay-Lac Saint Jean, Chicoutimi, Quebec

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Tripathy D, Blum JL, McCune S, Pluard T, Anderson D, Johnston A, Montelongo MZ, Zhang Z, Cappelleri JC, Gauthier E, Rocque GB. Real-world effectiveness of palbociclib plus hormone treatment and its impact on patient quality of life: a plain language summary of findings from POLARIS. Future Oncol. 2025 Nov;21(26):3359-3376. doi: 10.1080/14796694.2025.2570468. Epub 2025 Oct 27. PMID 41140056
- [Derived] Rocque GB, Blum JL, Ji Y, Pluard T, Migas J, Lakhanpal S, Jepsen E, Gauthier E, Wang Y, Montelongo MZ, Cappelleri JC, Chen C, Karuturi MS, Tripathy D. Enhancing the interpretation of real-world quality of life in patients with hormone receptor-positive/human epidermal growth factor receptor 2-negative advanced breast cancer enrolled in the POLARIS study. Oncologist. 2025 Oct 1;30(10):oyaf281. doi: 10.1093/oncolo/oyaf281. PMID 40971858
- [Derived] Tripathy D, Blum JL, Zhang H, Deng S, McCune SL, Patel K, Wang Y, Lakhanpal S, Karuturi MS, Zhang Z, Deshpande C, Montelongo MZ, Gauthier E, Liu Y, Rocque GB, Bardia A. Circulating Tumor DNA Genotyping of Intrinsic and Acquired Gene Alterations in Patients With Advanced Breast Cancer Receiving Palbociclib: Biomarker Results From POLARIS Study. JCO Precis Oncol. 2025 Aug;9:e2400810. doi: 10.1200/PO-24-00810. Epub 2025 Aug 18. PMID 40825169
- [Derived] Rocque GB, Blum JL, Ji Y, Pluard T, Migas J, Lakhanpal S, Jepsen E, Wang Y, Montelongo MZ, Zhang Z, Gauthier E, Tripathy D. Relationship of Prior Anticancer Treatments with Palbociclib Clinical Outcomes in Patients with HR+/HER2- Advanced Breast Cancer in Real-World Settings. Target Oncol. 2025 Jul;20(4):679-692. doi: 10.1007/s11523-025-01158-0. Epub 2025 Jun 24. PMID 40553419
- [Derived] Rocque GB, Blum JL, Ji Y, Pluard T, Migas J, Lakhanpal S, Jepsen E, Gauthier E, Wang Y, Montelongo MZ, Cappelleri JC, Karuturi MS, Tripathy D. Real-world quality-of-life of patients with HR+/HER2- advanced breast cancer treated with palbociclib plus endocrine therapy: EORTC QLQ-C30 results from POLARIS. Breast Cancer Res Treat. 2025 Feb;209(3):613-627. doi: 10.1007/s10549-024-07524-2. Epub 2024 Nov 25. PMID 39581892
- [Derived] Tripathy D, Blum JL, Karuturi MS, McCune S, Kurian S, Moezi M, Anderson D, Gauthier E, Zhang Z, Montelongo MZ, Wang Y, Rocque GB. Real-world effectiveness of palbociclib plus endocrine therapy in HR+/HER2- advanced breast cancer: final results from the POLARIS trial. Oncologist. 2025 Jul 4;30(7):oyae291. doi: 10.1093/oncolo/oyae291. PMID 39475418
- [Derived] Karuturi MS, Cappelleri JC, Blum JL, Patel K, Telivala B, McCune S, Cuevas JD, Lakhanpal S, Montelongo MZ, Wang Y, Tripathy D, Rocque GB. Measures of functional status in older patients treated with palbociclib for advanced breast cancer. J Geriatr Oncol. 2024 Jan;15(1):101670. doi: 10.1016/j.jgo.2023.101670. Epub 2023 Dec 6. PMID 38061288
- [Derived] Blum JL, DiCristo C, Gordon D, Karuturi MS, Oubre D, Jepsen E, Cuevas J, Lakhanpal S, Montelongo MZ, Zhang Z, Cappelleri JC, Wang Y, Tripathy D. Outcomes of male patients with HR+/HER2- advanced breast cancer receiving palbociclib in the real-world POLARIS study. Breast Cancer Res Treat. 2024 Feb;203(3):463-475. doi: 10.1007/s10549-023-07145-1. Epub 2023 Oct 30. PMID 37903899
- [Derived] Tripathy D, Blum JL, Rocque GB, Bardia A, Karuturi MS, Cappelleri JC, Liu Y, Zhang Z, Davis KL, Wang Y. POLARIS: a prospective, multicenter, noninterventional study assessing palbociclib in hormone receptor-positive advanced breast cancer. Future Oncol. 2020 Nov;16(31):2475-2485. doi: 10.2217/fon-2020-0573. Epub 2020 Aug 13. PMID 32787449
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481082

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with hormone receptor positive (HR+)/human epidermal growth factor receptor 2 negative (HER2-) advanced breast cancer (ABC) who were prescribed palbociclib in routine clinical practice across the United States and Canada were enrolled in this prospective observational study. Participants were followed up for approximately 3 years post end of treatment or until withdrawal from the study or death.
Pre-assignment Details: A total of 1285 participants were enrolled in the study. However, only 1250 participants initiated treatment with palbociclib.
Groups:
- Palbociclib + Endocrine Therapy: Participants with HR+/HER2- advanced breast cancer who were prescribed palbociclib in combination with endocrine treatment (Palbociclib, Fulvestrant, and Other) by the treating physician in routine clinical practice were included.
Period: Overall Study
Arm/Group | Palbociclib + Endocrine Therapy
Started | 1250
Completed | 54
Not Completed | 1196
Not completed — Death | 505
Not completed — Study terminated by sponsor | 383
Not completed — Other | 148
Not completed — No longer willing to participate in study | 101
Not completed — Lost to follow up | 39
Not completed — Adverse Event | 20

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all eligible participants enrolled in the study and received at least one dose of study medication.
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 1250
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.0 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1235
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 106
  Not Hispanic or Latino | 1106
  Unknown or Not Reported | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8
  Asian | 23
  Native Hawaiian or Other Pacific Islander | 5
  Black or African American | 139
  White | 1022
  More than one race | 0
  Unknown or Not Reported | 53

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants According to Real-World Tumor Response
Description: Real world tumor response included complete response (CR), Partial response (PR), Stable disease (SD), Progressive Disease (PD), and was determined by physician based on imaging, biopsies, biomarkers, and/or clinical judgment. Response as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) criteria may not be available for all participants. rwTR was derived as the best tumor response recorded from the palbociclib combination treatment start date until the first documentation of progressive disease. Only response assessments recorded on or before the start date of next subsequent line of treatment will be considered.
Time Frame: From start of palbociclib combination treatment until first documentation of progression (up to approximately 3 years)
Population: Safety analysis set included all participants enrolled in the study and received at least one dose of study medication. Here, 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 1250
Participants
  Overall: Complete response | 72
  Overall: Partial Response | 310
  Overall: Stable disease | 499
  Overall: Progressive disease | 223
  Overall: Indeterminate | 146
  1 Line of treatment: number analyzed (Participants) | 908
  1 Line of treatment: Complete response | 58
  1 Line of treatment: Partial Response | 248
  1 Line of treatment: Stable disease | 352
  1 Line of treatment: Progressive disease | 144
  1 Line of treatment: Indeterminate | 106
  2 or more lines of treatment: number analyzed (Participants) | 342
  2 or more lines of treatment: Complete response | 14
  2 or more lines of treatment: Partial Response | 62
  2 or more lines of treatment: Stable disease | 147
  2 or more lines of treatment: Progressive disease | 79
  2 or more lines of treatment: Indeterminate | 40

2. Primary Outcome: Real-World Tumor Response Rate
Description: Real world tumor response rate was defined as the percentage of participants with a best tumor response of complete response or partial response. Tumor response was determined by physician based on imaging, biopsies, biomarkers, and/or clinical judgment. RECIST criteria may not be available for all participants.
Time Frame: From start of palbociclib combination treatment until first documentation of progression (up to approximately 3 years)
Population: Safety analysis set included all participants who were enrolled in the study and received at least one dose of study medication. Here, 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 1250
Percentage of participants
  Overall | 30.6 [28.0 to 33.2]
  1 Line of treatment: number analyzed (Participants) | 908
  1 Line of treatment | 33.7 [30.6 to 36.9]
  2 or more lines of treatment: number analyzed (Participants) | 342
  2 or more lines of treatment | 22.2 [17.9 to 27.0]

3. Primary Outcome: Real World Progression Free Survival
Description: Real world progression free survival was defined as time (months) from initiation of the palbociclib combination treatment to the earliest of clinician-documented progression or death due to any cause, whichever occurred first. Participants without documented disease progression or death were censored at the last date of response assessment.
Time Frame: From initiation of the palbociclib combination treatment to the earliest of clinician-documented progression or death due to any cause, whichever occurs first. (up to approximately 3 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 1250
Months
  Overall | 18.8 [17.2 to 20.5]
  1 line of treatment: number analyzed (Participants) | 908
  1 line of treatment | 21.0 [18.8 to 24.7]
  2 or more lines of treatment: number analyzed (Participants) | 342
  2 or more lines of treatment | 13.2 [10.4 to 16.8]

4. Primary Outcome: Overall Survival
Description: Overall survival was defined as time from initiation of the palbociclib combination treatment to date of death due to any cause. Participants without a documented death were censored at last available visit date known to be alive.
Time Frame: From initiation of the palbociclib combination treatment to death due to any cause or censored, (up to approximately 3 years)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 1250
Months
  Overall | 42.3 [39.3 to 47.1]
  1 line of treatment: number analyzed (Participants) | 908
  1 line of treatment | 48.5 [42.0 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number participants with the events.
  2 or more lines of treatment: number analyzed (Participants) | 342
  2 or more lines of treatment | 37.2 [31.2 to 40.8]

5. Primary Outcome: Absolute Eastern Co-Operative Oncology Group (ECOG) Performance Status Scores at Baseline: Participants More Than or Equal to 70 Years Only
Description: ECOG performance status was a 6-level item used to assess the physical health of participants and ranged from 0 (fully active) to 5 (dead).
Time Frame: Baseline (last observed measurement prior to treatment start date)
Population: Safety analysis set included all participants who were enrolled in the study and received at least one dose of study medication. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 366
Units on a scale | 0.7 (0.74)

6. Primary Outcome: ECOG Performance Status Scores at Month 1: Participants More Than or Equal to 70 Years Only
Description: as for outcome 5
Time Frame: Month 1
Population: Safety analysis set included all participants who were enrolled in the study and received at least one dose of study medication, Here 'Overall Number of Participants Analyzed' signifies participants evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 326
Units on a scale | 0.7 (0.73)

7. Primary Outcome: ECOG Performance Status Scores at Month 2: Participants More Than or Equal to 70 Years Only
Description: as for outcome 5
Time Frame: Month 2
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 294
Units on a scale | 0.7 (0.70)

8. Primary Outcome: ECOG Performance Status Scores at Month 3: Participants More Than or Equal to 70 Years Only
Description: as for outcome 5
Time Frame: Month 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 297
Units on a scale | 0.7 (0.71)

9. Primary Outcome: ECOG Performance Status Scores at Month 6: Participants More Than or Equal to 70 Years Only
Description: as for outcome 5
Time Frame: Month 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 275
Units on a scale | 0.8 (0.73)

10. Primary Outcome: ECOG Performance Status Scores at Month 9: Participants More Than or Equal to 70 Years Only
Description: as for outcome 5
Time Frame: Month 9
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 224
Units on a scale | 0.8 (0.71)

11. Primary Outcome: ECOG Performance Status Scores at Month 12: Participants More Than or Equal to 70 Years Only
Description: as for outcome 5
Time Frame: Month 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 193
Units on a scale | 0.8 (0.75)

12. Primary Outcome: ECOG Performance Status Scores at Month 15: Participants More Than or Equal to 70 Years Only
Description: as for outcome 5
Time Frame: Month 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 165
Units on a scale | 0.8 (0.75)

13. Primary Outcome: ECOG Performance Status Scores at Month 18: Participants More Than or Equal to 70 Years Only
Description: as for outcome 5
Time Frame: Month 18
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 116
Units on a scale | 0.7 (0.74)

14. Primary Outcome: ECOG Performance Status Scores at Month 21: Participants More Than or Equal to 70 Years Only
Description: as for outcome 5
Time Frame: Month 21
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 80
Units on a scale | 0.8 (0.82)

15. Primary Outcome: ECOG Performance Status Scores at Month 24: Participants More Than or Equal to 70 Years Only
Description: as for outcome 5
Time Frame: Month 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 67
Units on a scale | 0.7 (0.81)

16. Primary Outcome: ECOG Performance Status Scores in Month 27: Participants More Than or Equal to 70 Years Only
Description: as for outcome 5
Time Frame: Month 27
Population: Safety analysis set included all participants who were enrolled in the study and received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 41
Units on a scale | 0.9 (0.88)

17. Primary Outcome: ECOG Performance Status Scores at Month 30: Participants More Than or Equal to 70 Years Only
Description: as for outcome 5
Time Frame: Month 30
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 25
Units on a scale | 0.9 (0.86)

18. Primary Outcome: ECOG Performance Status Scores at Month 33: Participants More Than or Equal to 70 Years Only
Description: as for outcome 5
Time Frame: Month 33
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 11
Units on a scale | 0.9 (0.70)

19. Primary Outcome: ECOG Performance Status Scores in Month 36: Participants More Than or Equal to 70 Years Only
Description: as for outcome 5
Time Frame: Month 36
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 7
Units on a scale | 0.6 (0.53)

20. Primary Outcome: ECOG Performance Status Scores at Month 39: Participants More Than or Equal to 70 Years Only
Description: as for outcome 5
Time Frame: Month 39
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 5
Units on a scale | 0.4 (0.55)

21. Primary Outcome: ECOG Performance Status Scores at Month 42: Participants More Than or Equal to 70 Years Only
Description: as for outcome 5
Time Frame: Month 42
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 2
Units on a scale | 0.5 (0.71)

22. Primary Outcome: Geriatric 8 Screening Tool Scores at Baseline: Participants More Than or Equal to 70 Years Only
Description: The G8 Screening Tool consisted of 7 items based on the Mini-Nutritional Assessment and a single item covering the participants age. Specifically, the G8 assessed food intake, weight changes, mobility, neuropsychological problems, body mass index, prescription count, and health status compared to similarly aged participants. Points were associated to each item and index score was calculated by summing points. The index score ranged in value from 0 (heavily impaired) to 17 (not at all impaired). If any of the 8 items was missing, the total score was missing.
Time Frame: Baseline (last observed measurement prior to treatment start date)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 354
Units on a scale | 13.4 (2.24)

23. Primary Outcome: Geriatric 8 Screening Tool Scores at Month 1: Participants More Than or Equal to 70 Years Only
Description: as for outcome 22
Time Frame: Month 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 300
Units on a scale | 13.3 (2.23)

24. Primary Outcome: Geriatric 8 Screening Tool Scores at Month 2: Participants More Than or Equal to 70 Years Only
Description: as for outcome 22
Time Frame: Month 2
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 255
Units on a scale | 13.4 (2.36)

25. Primary Outcome: Geriatric 8 Screening Tool Scores at Month 3: Participants More Than or Equal to 70 Years Only
Description: as for outcome 22
Time Frame: Month 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 180
Units on a scale | 13.4 (2.20)

26. Primary Outcome: Geriatric 8 Screening Tool Scores at Month 6: Participants More Than or Equal to 70 Years Only
Description: as for outcome 22
Time Frame: Month 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 215
Units on a scale | 13.5 (2.05)

27. Primary Outcome: Geriatric 8 Screening Tool Scores at Month 9: Participants More Than or Equal to 70 Years Only
Description: as for outcome 22
Time Frame: Month 9
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 181
Units on a scale | 13.7 (1.90)

28. Primary Outcome: Geriatric 8 Screening Tool Scores at Month 12: Participants More Than or Equal to 70 Years Only
Description: as for outcome 22
Time Frame: Month 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 137
Units on a scale | 13.7 (1.97)

29. Primary Outcome: Geriatric 8 Screening Tool Scores at Month 15: Participants More Than or Equal to 70 Years Only
Description: as for outcome 22
Time Frame: Month 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 104
Units on a scale | 13.6 (2.06)

30. Primary Outcome: Geriatric 8 Screening Tool Scores at Month 18: Participants More Than or Equal to 70 Years Only
Description: as for outcome 22
Time Frame: Month 18
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Palbociclib+ Endocrine Therapy: Participant with HR+/HER2- advanced breast cancer who were prescribed palbociclib in combination with other treatments by the treating physician in routine clinical practice were included.
Arm/Group | Palbociclib+ Endocrine Therapy
Number analyzed (Participants) | 83
Units on a scale | 13.4 (2.26)

31. Primary Outcome: Geriatric 8 Screening Tool Scores at Month 21: Participants More Than or Equal to 70 Years Only
Description: as for outcome 22
Time Frame: Month 21
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 55
Units on a scale | 13.4 (1.70)

32. Primary Outcome: Geriatric 8 Screening Tool Scores at Month 24: Participants More Than or Equal to 70 Years Only
Description: as for outcome 22
Time Frame: Month 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 44
Units on a scale | 13.5 (2.33)

33. Primary Outcome: Geriatric 8 Screening Tool Scores at Month 27: Participants More Than or Equal to 70 Years Only
Description: as for outcome 22
Time Frame: Month 27
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 28
Units on a scale | 13.3 (2.17)

34. Primary Outcome: Geriatric 8 Screening Tool Scores at Month 30: Participants More Than or Equal to 70 Years Only
Description: as for outcome 22
Time Frame: Month 30
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 16
Units on a scale | 13.1 (1.98)

35. Primary Outcome: Geriatric 8 Screening Tool Scores at Month 33: Participants More Than or Equal to 70 Years Only
Description: as for outcome 22
Time Frame: Month 33
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 13
Units on a scale | 13.3 (1.89)

36. Primary Outcome: Geriatric 8 Screening Tool Scores at Month 36: Participants More Than or Equal to 70 Years Only
Description: as for outcome 22
Time Frame: Month 36
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 4
Units on a scale | 14.1 (1.44)

37. Primary Outcome: Geriatric 8 Screening Tool Scores at Month 39: Participants More Than 70 or Equal to Years Only
Description: as for outcome 22
Time Frame: Month 39
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 4
Units on a scale | 13.5 (2.65)

38. Primary Outcome: Geriatric 8 Screening Tool Scores at Month 42: Participants More Than or Equal to 70 Years Only
Description: as for outcome 22
Time Frame: Month 42
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 2
Units on a scale | 13.0 (1.41)

39. Primary Outcome: Change From Baseline to Month 6 in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Scores at Baseline
Description: European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire 30: 30 item questionnaires composed of 5 functional subscales (physical, role, cognitive, emotional, and social); a global health/global quality of life scale; 3 symptom subscales (fatigue, pain and nausea/vomiting); and 6 single items that assessed additional symptoms (dyspnea, appetite loss, insomnia, constipation, diarrhea and financial difficulties). All scales and single item measures ranged in score from 0 to 100. Higher scores on functional and global quality of life scales represent better level of functioning. Higher scores on the symptom oriented scales represent more severe symptoms.
Time Frame: Baseline (last observed measurement prior to treatment start date) and Month 6
Population: Safety analysis set included all participants who were enrolled in the study and received at least one dose of study medication. All participants reported under 'Number of Participants Analyzed' contributed data to the table; however, may not have evaluable data for every row. Here 'Number Analyzed' signifies number of participants who provided an answer on the QoL Questionnaire for the specific item listed on each row.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 1250
Units on a scale
  Global health status/QoL: number analyzed (Participants) | 699
  Global health status/QoL | 3.5 (22.5)
  Dyspnoea: number analyzed (Participants) | 699
  Dyspnoea | -1.9 (27.7)
  Insomnia: number analyzed (Participants) | 701
  Insomnia | -0.9 (32.8)
  Appetite loss: number analyzed (Participants) | 702
  Appetite loss | -4.5 (31.3)
  Constipation: number analyzed (Participants) | 702
  Constipation | -1.7 (29.1)
  Diarrhoea: number analyzed (Participants) | 700
  Diarrhoea | 0.5 (24.8)
  Financial difficulties: number analyzed (Participants) | 700
  Financial difficulties | -0.7 (30.4)
  Physical functioning: number analyzed (Participants) | 702
  Physical functioning | 1.9 (19.3)
  Role functioning: number analyzed (Participants) | 702
  Role functioning | 4.2 (31.5)
  Emotional functioning: number analyzed (Participants) | 701
  Emotional functioning | 4.9 (20.3)
  Cognitive functioning: number analyzed (Participants) | 701
  Cognitive functioning | 0.6 (20.9)
  Social functioning: number analyzed (Participants) | 700
  Social functioning | 3.9 (27.2)
  Fatigue: number analyzed (Participants) | 702
  Fatigue | -0.7 (25.0)
  Nausea and vomiting: number analyzed (Participants) | 702
  Nausea and vomiting | -1.7 (20.9)
  Pain: number analyzed (Participants) | 702
  Pain | -6.9 (29.8)

40. Primary Outcome: Change From Baseline to Month 12 in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Scores at Baseline
Description: EORTC QLQ-C30: 30 item questionnaire composed of 5 functional subscales (physical, role, cognitive, emotional, and social); a global health/global quality of life scale; 3 symptom subscales (fatigue, pain and nausea/vomiting); and 6 single items that assessed additional symptoms (dyspnea, appetite loss, insomnia, constipation, diarrhea and financial difficulties). All scales and single item measures ranged in score from 0 to 100. Higher scores on functional and global quality of life scales represent better level of functioning. Higher scores on the symptom oriented scales represent more severe symptoms.
Time Frame: Baseline (last observed measurement prior to treatment start date) and Month 12
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 1250
Units on a scale
  Global health status/QoL: number analyzed (Participants) | 466
  Global health status/QoL | 2.5 (23.1)
  Dyspnoea: number analyzed (Participants) | 465
  Dyspnoea | -1.8 (29.3)
  Insomnia: number analyzed (Participants) | 466
  Insomnia | -3.1 (32.9)
  Appetite loss: number analyzed (Participants) | 467
  Appetite loss | -5.1 (32.1)
  Constipation: number analyzed (Participants) | 467
  Constipation | -1.9 (26.3)
  Diarrhoea: number analyzed (Participants) | 465
  Diarrhoea | 0.1 (23.5)
  Financial difficulties: number analyzed (Participants) | 464
  Financial difficulties | -3.1 (28.9)
  Physical functioning: number analyzed (Participants) | 467
  Physical functioning | 1.2 (20.0)
  Role functioning: number analyzed (Participants) | 467
  Role functioning | 4.5 (32.3)
  Emotional functioning: number analyzed (Participants) | 466
  Emotional functioning | 4.7 (20.4)
  Cognitive functioning: number analyzed (Participants) | 466
  Cognitive functioning | 0.1 (21.5)
  Social functioning: number analyzed (Participants) | 466
  Social functioning | 3.4 (29.0)
  Fatigue: number analyzed (Participants) | 467
  Fatigue | -0.4 (25.9)
  Nausea and vomiting: number analyzed (Participants) | 467
  Nausea and vomiting | -1.3 (21.2)
  Pain: number analyzed (Participants) | 467
  Pain | -5.7 (30.2)

41. Primary Outcome: Change From Baseline to Month 18 in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Scores at Baseline
Description: as for outcome 40
Time Frame: Baseline (last observed measurement prior to treatment start date) and Month 18
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 1250
Units on a scale
  Global health status/QoL: number analyzed (Participants) | 338
  Global health status/QoL | 2.5 (24.5)
  Dyspnoea: number analyzed (Participants) | 339
  Dyspnoea | 0.4 (28.3)
  Insomnia: number analyzed (Participants) | 339
  Insomnia | -3.5 (32.8)
  Appetite loss: number analyzed (Participants) | 339
  Appetite loss | -4.7 (31.7)
  Constipation: number analyzed (Participants) | 339
  Constipation | -1.4 (30.3)
  Diarrhoea: number analyzed (Participants) | 335
  Diarrhoea | 0.8 (26.9)
  Financial difficulties: number analyzed (Participants) | 338
  Financial difficulties | -2.5 (30.9)
  Physical functioning: number analyzed (Participants) | 340
  Physical functioning | 1.6 (21.6)
  Role functioning: number analyzed (Participants) | 340
  Role functioning | 6.0 (33.7)
  Emotional functioning: number analyzed (Participants) | 339
  Emotional functioning | 5.9 (19.4)
  Cognitive functioning: number analyzed (Participants) | 339
  Cognitive functioning | -0.9 (22.2)
  Social functioning: number analyzed (Participants) | 339
  Social functioning | 4.8 (28.9)
  Fatigue: number analyzed (Participants) | 339
  Fatigue | -1.8 (26.0)
  Nausea and vomiting: number analyzed (Participants) | 340
  Nausea and vomiting | -2.2 (22.1)
  Pain: number analyzed (Participants) | 340
  Pain | -7.6 (31.8)

42. Primary Outcome: Activities of Daily Living Scores at Baseline: Participants More Than or Equal to 70 Years Only
Description: Activities of Daily Living is assessed using a six-item ADL limitations measure that inventoried whether participants had difficulty bathing, dressing, toileting, feeding, with transfer, and incontinence. Each item was rated on a 3-point Likert scale measuring independence in performing the activity and scores ranged from 1 to 3; where, 1=unable to do without assistance, 2=partial assistance needed and 3=no assistance. The total score was calculated as a sum of scores of individual items and ranged between 6 to 18, where a score of 6 indicated a very dependent participant and a score of 18 represented an independent participant.
Time Frame: Baseline (last observed measurement prior to treatment start date)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 365
Units on a scale | 17.6 (1.14)

43. Primary Outcome: Activities of Daily Living Scores at Month 1: Participants More Than or Equal to 70 Years Only
Description: Activities of Daily Living is assessed using a six-item ADL limitations measure that inventoried whether participants had difficulty bathing, dressing, toileting, feeding, with transfer, and incontinence. Each item was rated on a 3-point Likert scale measuring independence in performing the activity and scores ranged from 1 to 3; where, 1=unable to do without assistance, 2=partial assistance needed and 3=no assistance. The total score was calculated as a sum of scores of individual items and ranged between 6 to 18, where a score of 6 indicated a very dependent participant and a score of 18 represented an independent participants.
Time Frame: Month 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 313
Units on a scale | 17.6 (1.23)

44. Primary Outcome: Activities of Daily Living Scores at Month 2: Participants More Than or Equal to 70 Years Only
Description: as for outcome 43
Time Frame: Month 2
Population: Safety analysis set included all participants who were enrolled in the study and received at least one dose of study medication, 'Overall Number of Participants Analyzed' signifies participants evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 269
Units on a scale | 17.7 (1.08)

45. Primary Outcome: Activities of Daily Living Scores at Month 3: Participants More Than or Equal to 70 Years Only
Description: as for outcome 43
Time Frame: Month 3
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 193
Units on a scale | 17.6 (1.00)

46. Primary Outcome: Activities of Daily Living Scores Month 6: Participants More Than or Equal to 70 Years Only
Description: as for outcome 43
Time Frame: Month 6
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 228
Units on a scale | 17.6 (1.19)

47. Primary Outcome: Activities of Daily Living Scores at Month 9: Participants More Than or Equal to 70 Years Only
Description: as for outcome 43
Time Frame: Month 9
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 185
Units on a scale | 17.6 (1.47)

48. Primary Outcome: Activities of Daily Living Scores at Month 12: Participants More Than or Equal to 70 Years Only
Description: as for outcome 43
Time Frame: Month 12
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 140
Units on a scale | 17.4 (1.55)

49. Primary Outcome: Activities of Daily Living Scores at Month 15: Participants More Than or Equal to 70 Years Only
Description: as for outcome 43
Time Frame: Month 15
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 112
Units on a scale | 17.5 (1.52)

50. Primary Outcome: Activities of Daily Living Scores at Month 18: Participants More Than or Equal to 70 Years Only
Description: as for outcome 42
Time Frame: Month 18
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 85
Units on a scale | 17.6 (1.13)

51. Primary Outcome: Activities of Daily Living Scores at Month 21: Participants More Than or Equal to 70 Years Only
Description: as for outcome 43
Time Frame: Month 21
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 57
Units on a scale | 17.7 (0.91)

52. Primary Outcome: Activities of Daily Living Scores at Month 24: Participants More Than or Equal to 70 Years Only
Description: as for outcome 43
Time Frame: Month 24
Population: Safety analysis set included all participants who were enrolled in the study and received at least one dose of study medication.'Overall Number of Participants Analyzed' signifies participants evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 48
Units on a scale | 17.6 (0.93)

53. Primary Outcome: Activities of Daily Living Scores at Month 27: Participants More Than or Equal to 70 Years Only
Description: as for outcome 43
Time Frame: Month 27
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 27
Units on a scale | 17.5 (1.01)

54. Primary Outcome: Activities of Daily Living Scores at Month 30: Participants More Than or Equal to 70 Years Only
Description: as for outcome 43
Time Frame: Month 30
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 16
Units on a scale | 17.3 (2.05)

55. Primary Outcome: Activities of Daily Living Scores at Month 33: Participants More Than or Equal to 70 Years Only
Description: as for outcome 43
Time Frame: Month 33
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 13
Units on a scale | 17.5 (1.66)

56. Primary Outcome: Activities of Daily Living Scores at Month 36: Participants More Than or Equal to 70 Years Only
Description: as for outcome 43
Time Frame: Month 36
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 4
Units on a scale | 17.3 (1.50)

57. Primary Outcome: Activities of Daily Living Scores at Month 39: Participants More Than or Equal to 70 Years Only
Description: as for outcome 43
Time Frame: Month 39
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 4
Units on a scale | 17.3 (1.50)

58. Primary Outcome: Activities of Daily Living Scores at Month 42: Participants More Than or Equal to 70 Years Only
Description: as for outcome 43
Time Frame: Month 42
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 2
Units on a scale | 16.5 (2.12)

59. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in administered medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage.
Time Frame: From start of palbociclib treatment or date of informed consent until 28 days after last dose of study treatment (up to approximately 3 years)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Groups:
- Palbociclib+ Endocrine Therapy: Participants with HR+/HER2- advanced breast cancer who were prescribed palbociclib in combination with endocrine treatment (Palbociclib, Fulvestrant, and Other) by the treating physician in routine clinical practice were included.
Arm/Group | Palbociclib+ Endocrine Therapy
Number analyzed (Participants) | 1250
Participants | 1123

60. Primary Outcome: Number of Participants With Serious Adverse Events
Description: A serious adverse event was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) at any dose that: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); resulted in congenital anomaly/birth defect.
Time Frame: as for outcome 59
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib+ Endocrine Therapy
Number analyzed (Participants) | 1250
Participants | 403

61. Primary Outcome: Number of Participants With Any Clinical Laboratory Abnormalities
Description: Following lab parameters were assessed Anemia, Hemoglobin increased, Lymphocyte count decreased, Lymphocyte count increased, Neutrophil count decreased, Platelet count decreased, Leukocyte count decreased, Leukocyte count increased, Number of participants with any lab abnormality was reported.
Time Frame: as for outcome 59
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Endocrine Therapy
Number analyzed (Participants) | 1250
Participants | 1170

ADVERSE EVENTS:
Time Frame: From start of palbociclib treatment or date of informed consent until 28 days after last dose of study treatment (up to approximately 3 years)
Description: Same event may appear as both non-SAE and SAE. What is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in other participant, or a participant may have experienced both SAE and non-SAE. Safety analysis set included all participants enrolled in the study and received at least one dose of study medication.
Arm/Group | Palbociclib + Endocrine Therapy
All-Cause Mortality (participants affected / at risk) | 505/1250
Serious Adverse Events (participants affected / at risk) | 403/1250
Other Adverse Events (participants affected / at risk) | 1035/1250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib + Endocrine Therapy (N=1250)
Neutropenia (Blood and lymphatic system disorders) | 4
Anaemia (Blood and lymphatic system disorders) | 18
Leukopenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 8
Pancytopenia (Blood and lymphatic system disorders) | 3
Leukocytosis (Blood and lymphatic system disorders) | 1
Neutrophil count decreased (Investigations) | 5
White blood cell count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 5
Transaminases increased (Investigations) | 2
Blood creatinine increased (Investigations) | 1
Blood creatine increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Respiratory syncytial virus test positive (Investigations) | 1
Weight decreased (Investigations) | 1
Sepsis (Infections and infestations) | 22
Pneumonia (Infections and infestations) | 20
Urinary tract infection (Infections and infestations) | 15
Cellulitis (Infections and infestations) | 9
Septic shock (Infections and infestations) | 3
Appendicitis (Infections and infestations) | 4
Influenza (Infections and infestations) | 4
Bronchitis (Infections and infestations) | 2
Diverticulitis (Infections and infestations) | 3
Kidney infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Abscess (Infections and infestations) | 2
Bacteraemia (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 2
Empyema (Infections and infestations) | 2
Postoperative wound infection (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 2
Urosepsis (Infections and infestations) | 2
Beta haemolytic streptococcal infection (Infections and infestations) | 1
Breast cellulitis (Infections and infestations) | 1
Corona virus infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Neutropenic sepsis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Pneumonia viral (Infections and infestations) | 1
Post procedural infection (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Disease progression (General disorders) | 36
Fatigue (General disorders) | 2
Asthenia (General disorders) | 12
Death (General disorders) | 7
Pain (General disorders) | 2
Chest pain (General disorders) | 6
Pyrexia (General disorders) | 8
Oedema peripheral (General disorders) | 3
Non-cardiac chest pain (General disorders) | 2
Hernia obstructive (General disorders) | 1
Systemic inflammatory response syndrome (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 12
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 13
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 20
Vomiting (Gastrointestinal disorders) | 24
Diarrhoea (Gastrointestinal disorders) | 9
Abdominal pain (Gastrointestinal disorders) | 10
Small intestinal obstruction (Gastrointestinal disorders) | 9
Ascites (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 3
Intestinal obstruction (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 3
Colitis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Obstruction gastric (Gastrointestinal disorders) | 2
Oesophagitis (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Enteritis (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Intestinal perforation (Gastrointestinal disorders) | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1
Peptic ulcer (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 23
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Inflammatory carcinoma of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 11
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 7
Decreased appetite (Metabolism and nutrition disorders) | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2
Failure to thrive (Metabolism and nutrition disorders) | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1
Syncope (Nervous system disorders) | 5
Headache (Nervous system disorders) | 5
Cerebrovascular accident (Nervous system disorders) | 8
Ischaemic stroke (Nervous system disorders) | 2
Metabolic encephalopathy (Nervous system disorders) | 3
Aphasia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Encephalopathy (Nervous system disorders) | 2
Brain oedema (Nervous system disorders) | 1
Cerebral artery occlusion (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cerebrovascular disorder (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Cardiac arrest (Cardiac disorders) | 7
Atrial fibrillation (Cardiac disorders) | 10
Cardiac failure congestive (Cardiac disorders) | 8
Acute myocardial infarction (Cardiac disorders) | 3
Pericardial effusion (Cardiac disorders) | 3
Angina pectoris (Cardiac disorders) | 3
Cardiomyopathy (Cardiac disorders) | 2
Arrhythmia (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Cardiac failure chronic (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Chronic left ventricular failure (Cardiac disorders) | 1
Left ventricular failure (Cardiac disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 1
Fall (Injury, poisoning and procedural complications) | 9
Hip fracture (Injury, poisoning and procedural complications) | 4
Femur fracture (Injury, poisoning and procedural complications) | 2
Humerus fracture (Injury, poisoning and procedural complications) | 2
fracture (Injury, poisoning and procedural complications) | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 2
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Compression fracture (Injury, poisoning and procedural complications) | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Acute kidney injury (Renal and urinary disorders) | 16
Hydronephrosis (Renal and urinary disorders) | 4
Nephrolithiasis (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal tubular necrosis (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Depression (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 3
Mental status changes (Psychiatric disorders) | 5
Hallucination (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Substance abuse (Psychiatric disorders) | 1
Hypotension (Vascular disorders) | 3
Deep vein thrombosis (Vascular disorders) | 3
Lymphoedema (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Hypovolaemic shock (Vascular disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 1
Vena cava thrombosis (Vascular disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 4
Acute hepatic failure (Hepatobiliary disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Diplopia (Eye disorders) | 1
Exophthalmos (Eye disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus arrest (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 3
Chest discomfort (General disorders) | 1
Medical device site joint infection (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Occult blood positive (Investigations) | 1
Haemorrhage intracranial (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Lacunar infarction (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 66
Cardiac Failure (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib + Endocrine Therapy (N=1250)
Neutropenia (Blood and lymphatic system disorders) | 415
Anaemia (Blood and lymphatic system disorders) | 310
Thrombocytopenia (Blood and lymphatic system disorders) | 112
Nausea (Gastrointestinal disorders) | 308
Diarrhoea (Gastrointestinal disorders) | 233
Constipation (Gastrointestinal disorders) | 133
Vomiting (Gastrointestinal disorders) | 117
Stomatitis (Gastrointestinal disorders) | 102
Fatigue (General disorders) | 444
White blood cell count decreased (Investigations) | 272
Neutrophil count decreased (Investigations) | 284
Platelet count decreased (Investigations) | 161
Lymphocyte count decreased (Investigations) | 116
Arthralgia (Musculoskeletal and connective tissue disorders) | 202
Back pain (Musculoskeletal and connective tissue disorders) | 150
Pain in extremity (Musculoskeletal and connective tissue disorders) | 89
Headache (Nervous system disorders) | 128
Dizziness (Nervous system disorders) | 105
Neuropathy peripheral (Nervous system disorders) | 68
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 125
Cough (Respiratory, thoracic and mediastinal disorders) | 107
Alopecia (Skin and subcutaneous tissue disorders) | 113
Hot flush (Vascular disorders) | 123
Decreased appetite (Metabolism and nutrition disorders) | 123
Insomnia (Psychiatric disorders) | 95
Urinary tract infection (Infections and infestations) | 78
Leukopenia (Blood and lymphatic system disorders) | 66
Aspartate aminotransferase increased (Investigations) | 66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-08-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT03280303/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT03280303/SAP_001.pdf